CLINICAL TRIAL: NCT03447483
Title: Cohort Study: Modelling Toxicity Processing in Patients Treated by Immunotherapy (MOTIVATE).
Acronym: MOTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17GENE22
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumor
Keywords: Solid tumor; Immune Checkpoint Inhibitor; immune-related Adverse Event

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of patients starting a treatment by ICI (Other)
  Interventions: Other: Patients starting a treatment by ICI

INTERVENTIONS:
Other: Patients starting a treatment by ICI — Completion of the Quality of Life Questionnaire Core 30 (QLQ-C30) before treatment administration and during the 12 months of treatment period, at the following time points:
  * every 6 weeks for treatment regimen administered every 2 or 3 weeks
  * at Weeks 6, 12, 20, 24 for treatment regimen administered every 4 weeks

SUMMARY:
This trial is a multicentric, prospective cohort study of 150 patients aiming to model evolution of toxicity over time in patients with solid tumor and starting first cycle of Immune Checkpoint Inhibitor (ICI) treatment.

The study will be conducted on a population of patients treated with ICI in the context of routine care. The follow-up during the treatment period and the clinical, biological and radiological assessments will be performed according to the standard of each centre.

The study data (immune-related adverse events) will be collected during each administration of the treatment.

A questionnaire will be completed by the patient before the treatment administrations.

Patients will be followed until disease progression or up to 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years old
2. Patient with a solid tumor whatever the organ
3. Patient receiving an Immune Checkpoint Inhibitor treatment
4. Patient starting first cycle of Immune Checkpoint Inhibitor treatment whatever the treatment line
5. Patient affiliated to the french social security system
6. Patient must provide written informed consent prior to inclusion in the study and any study-specific procedure

Exclusion Criteria:

1. Patient who must receive a treatment other than Immune Checkpoint Inhibitor
2. Patient with contraindication to the use of a checkpoint inhibitor (e.g., auto immune disorders requiring an immunosuppressive therapy)
3. Pregnant or breastfeeding women
4. Any psychological, familial, geographical or sociological condition potentially preventing the medical follow-up and/or study procedures
5. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of toxicities evaluated according to the classification of the Common for Toxicity Criteria for Adverse Events (CTCAE) V4.03 | 12 months by patient

SECONDARY OUTCOMES:
Time to appearance of toxicity | 12 months by patient
Rate of patients for which treatment was restarted among those who had stopped treatment for the management of an immune-related Adverse Event (irAE) | 12 months by patient
Quality of life using the QLQ-C30 questionnaire | 12 months by patient

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH ALBI, Albi
  - Ch Castres, Castres
  - Institut Regional Du Cancer de Montpellier (Icm), Montpellier
  - Institut Curie, Paris
  - Hopital Larrey, Toulouse
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse

REFERENCES:
- [Derived] Cabarrou B, Gomez-Roca C, Viala M, Rabeau A, Paulon R, Loirat D, Munsch N, Delord JP, Filleron T. Modernizing adverse events analysis in oncology clinical trials using alternative approaches: rationale and design of the MOTIVATE trial. Invest New Drugs. 2020 Dec;38(6):1879-1887. doi: 10.1007/s10637-020-00938-x. Epub 2020 May 7. PMID 32383099